CLINICAL TRIAL: NCT00634829
Title: Randomized, Double-Blind, Controlled, Single-Dose, Three-Treatment, Cross-Over Study of The Protective Effects Of Albuterol-HFA In Preventing Exercise-Induced Bronchoconstriction In Adolescent And Adult Asthmatic Patients
Brief Title: Single-Dose Cross-Over Study of the Effects of Albuterol-HFA in Exercise Induced Bronchoconstriction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: IND voluntarily withdrawn, without prejudice
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: API-A004-CLN-D
Record Dates: First submitted 2008-03-07; First posted 2008-03-13 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Asthma; Bronchospasm
MeSH Terms: conditions — Asthma; Bronchial Spasm | interventions — Albuterol; RNA aptamer SUP-A-004

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- T (Experimental): Armstrong Albuterol HFA Inhalation Aerosol
  Interventions: Drug: albuterol (Armstrong Albuterol HFA)
- R (Active Comparator): 2 inhalations Proventil-HFA Albuterol Sulfate, 108 mcg, prior to exercise
  Interventions: Drug: Albuterol Sulfate (Provenetil-HFA)
- P (Placebo Comparator): Placebo-HFA
  Interventions: Drug: Placebo-HFA

INTERVENTIONS:
Drug: albuterol (Armstrong Albuterol HFA) — 2 inhalations of 108 mcg albuterol sulfate prior to exercise, single dose
  Other Names: A004; Albuterol-HFA Inhalation Aerosol
  Arms: T
Drug: Albuterol Sulfate (Provenetil-HFA) — 2 inhalations of Proventil-HFA, 108 mcg/inhalation prior to exercise
  Other Names: Provenetil-HFA; albuterol sulfate-HFA
  Arms: R
Drug: Placebo-HFA — Placebo containing HFA propellant without active drug substance
  Arms: P

SUMMARY:
This clinical study will evaluate and establish the protective effects of Amphastar's Albuterol Sulfate HFA Inhalation Aerosol (Albuterol-HFA), in preventing exercise-induced bronchoconstriction (EIB) in adolescent and adult asthmatic patients, in comparison with (1) Proventil®-HFA (Reference drug and Active Control ), and (2) Placebo-HFA control (HFA propellant only). Safety of the test drug, Albuterol-HFA, will also be evaluated in comparison to the Active and Placebo Controls. Analyses will be performed to determine if the Armstrong's Albuterol-HFA has resulted in a significant bronchoprotective effect, with attenuated Max % Fall in FEV1, in comparison to the Placebo-HFA control.

DETAILED DESCRIPTION:
The prevalence of exercise-induced bronchoconstriction (EIB) has been reported to be around 70% to 75% among patients with clinically established asthma. Airway cooling and drying are thought to cause the release of inflammatory mediators, such as histamine and leukotrienes, which then mediate clinical EIB symptoms. Pretreatment with a variety of medications will ameliorate EIB. Albuterol has been found to be more effective in minimizing EIB than theophylline, ipratropiom, cromoglycate, etc. Tested using a treadmill exercise challenge, the newer formulations of albuterol MDI with HFA as propellant have been demonstrated to be as effective as those with CFC as propellant in protecting asthma patients from EIB in children and adults.

As a part of the Amphastar Pharmaceuticals' clinical development plan, the current study examines the clinical efficacy of A004, Armstrong Pharmaceuticals' Albuterol HFA oral inhalation MDI, in preventing EIB in adolescent and adult asthmatic patients.

This is a randomized, double-blind, active and placebo-controlled, three-treatment, cross-over study, to be conducted in adolescent and adult patients with mild to moderate asthma and demonstrable EIB.

All subjects will be screened against the inclusion/exclusion criteria for enrollment. A computer-generated randomization code will be created by the Amphastar Pharmaceuticals' IT Department, so that each enrolled subject will receive all three double-blinded treatments in randomized sequence. Each treatment is followed by a standardized exercise challenge and a series of FEV1 measurements during the 90 min post-exercise period. The three crossover Treatment Arms are:

* Treatment T (Armstrong's Test Drug: Albuterol-HFA);
* Treatment R (Reference Drug and Active Control: Proventil®-HFA);
* Treatment P (Placebo-HFA).

By the definition of the crossover design, the three Treatment Arms are expected to consist comparably of 24 evaluable subjects. The consecutive study sessions will be separated by an interval of 1-14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, aged 12 - 50 years, and in general good health.
2. A documented history of mild to moderate asthma, for at-least 6-months, requiring inhaled B-adrenergic agonists for symptom control.
3. Having a history of exercise-induced bronchoconstriction, that can be prevented or relieved by the use of an inhaled B-agonist.
4. Satisfying asthma stability requirement, such that over the 30 days prior to the screening, there are no significant changes in asthma therapy and no asthma-related hospitalization or emergency medical visits.
5. Being able to withhold treatment with inhaled bronchodilators and/or restricted medications for the minimum washout periods indicated in Appendix II prior to pulmonary function testing at Screening Visit and Clinical Visits 1, 2 and 3.
6. Having a baseline forced expiratory volume in the 1st second (FEV1) that is greater than nor equal to 65.0% of predicted normal values.
7. Demonstrating a greater than or equal to 20.0%, but <50.0%, fall in FEV1 during a Standard Exercise Challenge test per current ATS guidance, at Screening.
8. Demonstrating satisfactory techniques in the correct use of metered-dose inhaler (MDIs).
9. Female patients of child-bearing potential being non-pregnant and non-lactating, and using an acceptable method of contraception.
10. Willingness and ability to sign the informed consent and HIPPA forms to participate in this trial.

Exclusion Criteria:

1. A smoking history of ≥10 pack-years, or having smoked within the past 12 months prior to Screening.
2. Any current or past significant respiratory diseases that might significantly interfere with pharmacodynamic response to the study drugs, such as cystic fibrosis, bronchiectasis, emphysema, pulmonary malignancies, etc, other than asthma.
3. Clinically significant cardiovascular, hematological, renal, neurologic, hepatic, and endocrine disorders, or psychiatric diseases, or any other significant health conditions that in the opinion of the investigator might interfere with bronchodilator responses.
4. Recent upper or lower respiratory tract infection (within 4 weeks) prior to Screening.
5. Recent (per Appendix II, Part I) use of orally ingested or systemically administered corticosteroids, B-adrenergic bronchodilators, monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants (TCAs), B-blockers, or drugs that affect study drug performance.
6. Taking >1,000 mcg daily of inhaled beclomethasone dipropionate or budesonide, or >500 mcg daily of inhaled fluticasone propionate, or taking high doses of other orally inhaled corticosteroids that suggest severe asthma state, in the opinion of the investigator, within four weeks of Screening.
7. Demonstrating clinically significant abnormal 12-lead ECG results, upon Screening.
8. Any significant physical (e.g., musculoskeletal, overweight, etc) conditions that, in the opinion of the investigator, could limit the subject's ability to perform the exercise challenge test.
9. Known intolerance or hypersensitivity to any component of the MDI formulation (albuterol, HFA-134a, oleic acid and alcohol).
10. Known or reasonably suspected substance abuses.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The maximum percentage fall in FEV1, from the Pre-Exercise FEV1, between Albuterol-HFA and Placebo-HFA. | 90 minutes post exercise

SECONDARY OUTCOMES:
Evaluation of relative broncho-protective efficacy of Albuterol-HFA, in comparison to the active comparator, Proventil®-HFA, using the Max % fall in Post-Exercise FEV1, from the Pre-exercise FEV1 | 90 minutes post exercise
Pre-exercise FEV1 values (volume in Liters, recorded ), indicative of bronchodilator responsiveness. | 20-30 min post dose
Number and percentage of subjects who demonstrate a <20.0% fall in FEV1, from the Pre-exercise FEV1. | 90 min post-exercise
Area Under-the-Curve of percentage fall in FEV1, from the Pre-exercise FEV1. | 90 min post-exercise
Time to recovery, as the time point where FEV1 recovers from maximum percent fall in FEV1 to be within 5.0% of the Pre-Exercise FEV1 values. | concurrent with study visit
Number of subjects who cannot complete the exercise at specified intensity and length, due to asthma symptoms. | concurrent with study visit
Number of subjects requiring B2-agonist rescue inhalations during exercise, and during the 90 min post-exercise period. | 90 minutes post exercise
The following baseline and post-dose safety parameters before and after each exercise-challenge tests will be assessed: Vital signs: blood pressure (SBP/DBP) and heart rate (HR). | concurrent with study visit
12-lead ECG: HR, QT and QTc intervals, before and after treatment with Albuterol-HFA, versus the active control, and placebo control. | concurrent with study visit
Pre-study (Screening) and End-of-Study laboratory tests for CBC, blood chemistry panel, urinalysis and urine pregnancy test. | Throughout study
Adverse events and side effects will be documented when observed by investigators or reported by subjects. | throughout study

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Colorado Allergy and Asthma Center, Denver, Colorado
  - Colorado Allergy and Asthma Center, Englewood, Colorado
  - Colorado Allergy and Asthma Center, Lakewood, Colorado